CLINICAL TRIAL: NCT01572064
Title: Magnetic Resonance Imaging in the Evaluation of Hepatic Fibrosis: Search for MRI Biomarker
Brief Title: Magnetic Resonance Imaging in the Evaluation of Liver Fibrosis
Acronym: Mrker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 09/H0403/1
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Liver Fibrosis
Keywords: MRI; liver biopsy; serological markers
MeSH Terms: conditions — Liver Cirrhosis | interventions — Blood Specimen Collection; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood sample — 1 fasted blood sample taken for metabolomics
Other: MRI Scan — 1 single visit for MRI and MRS

SUMMARY:
The main purpose of this pilot study is to evaluate non-invasive magnetic resonance imaging (MRI) techniques in the detection and grading of liver fibrosis, so that the investigators can reduce the need of invasive techniques such as liver biopsy and transjugular hepatic venous portal pressure gradient (HVPG) measurements to assess the degree of liver scarring and portal hypertension.

DETAILED DESCRIPTION:
In chronic liver diseases of all aetiology, persistent hepatocyte injury leads to progressive fibrosis and cirrhosis. In the UK, 76 adults per 100,000 population have cirrhosis and its incidence is increasing (Fleming et al., J Hepatol 2008,49,p732-738). Currently, liver biopsy is the only method of assessing the degree of fibrosis. However, liver biopsy is associated with limitations such as sampling error, intra- and inter-observer variations in interpretation and adverse events (Morbidity 1-5% and mortality between 1 in 1,000 to 1 in 10,000), hence considered a 'Silver (rather than Gold) standard'. Assessment of degree of fibrosis is necessary to stage the disease process, determine the timing of intervention and for prognosis.

Development of portal hypertension as a result of progressive fibrosis is a landmark in the natural history of chronic liver diseases as it accounts for majority of complications and clinical outcome. The degree of fibrosis and presence of portal hypertension will determine whether patients are included in surveillance programmes for the early detection of varices and hepatocellular carcinoma. As with assessment of the degree of fibrosis, the presence and degree of portal hypertension can only be determined by transjugular hepatic venous portal pressure gradient (HVPG) measurements, another investigation that is also hampered by access, costs, risks and difficulty of serial measurements.

A variety of evolving techniques using magnetic resonance imaging (MRI) (Talwalkar et al., Hepatology 2008; 47:332-42) if validated and established, have potential to replace liver biopsy and HVPG measurements. The non-invasive nature of MRI, its ability to estimate amount of accumulated fat (1H MR spectroscopy), cell membrane turnover (31P-MRS), iron (relaxometry), fibrosis (MR elastography) as well as an ability to assess portal blood flow and hepatic perfusion (Arterial Spin Labelling (ASL)) make it an ideal tool to evaluate liver structure and function and to stage the liver disease. Most recently, MRI has seen unprecedented developments in terms of accuracy of quantitation and speed of assessment, which has been realised due to data-sharing ultra-fast MRI sequences, multispectral analysis, and refinement of elastography methods. Validation of evolving MRI techniques against liver biopsies, HVPG and metabolomics is a critical step prior to its translation into clinical applications by the creation of MRI biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Liver biopsy within the last 3 months
* Underlying chronic liver disease- hepatitis C, alcoholic liver disease, non-alcoholic fatty liver disease, hepatitis B, haemochromatosis or where biopsy is considered normal.
* Ability to consent to participate in the study

Exclusion Criteria:

* Inadequate biopsy length for histology
* Absolute contraindications for MRI
* Abdominal/waist circumference greater than 112 cm (44 inches), due to scanner bore constraints
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of MRI in the detection of fibrosis and advanced fibrosis compared with histology. | MRI within 3 months of liver biopsy
  MRI and MRS

SECONDARY OUTCOMES:
Diagnostic accuracy of MRI in the detection of fibrosis and advanced fibrosis compared with serological markers. | Blood Test taken on same day as MRI
  Metabolomics analysis

CONTACTS AND LOCATIONS:
Overall Officials: Guruprasad P Aithal, PhD, Principal Investigator — University of Nottingham
Locations (1):
- NDDC BRU and Sir Peter Mansfield Magnetic Resonance Centre, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Background] Talwalkar JA, Yin M, Fidler JL, Sanderson SO, Kamath PS, Ehman RL. Magnetic resonance imaging of hepatic fibrosis: emerging clinical applications. Hepatology. 2008 Jan;47(1):332-42. doi: 10.1002/hep.21972. PMID 18161879
- [Background] Fleming KM, Aithal GP, Solaymani-Dodaran M, Card TR, West J. Incidence and prevalence of cirrhosis in the United Kingdom, 1992-2001: a general population-based study. J Hepatol. 2008 Nov;49(5):732-8. doi: 10.1016/j.jhep.2008.05.023. Epub 2008 Jun 25. PMID 18667256